CLINICAL TRIAL: NCT01923272
Title: Non-Invasive Neurostimulation of the Vagus Nerve With the AlphaCore Device for the Relief of Exercised Induced Bronchoconstriction
Brief Title: Non-Invasive Neurostimulation of the Vagus Nerve With the AlphaCore Device for the Relief of EIB
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Similar study being conducted, Sponsor decided to not duplicate study
Sponsor: ElectroCore INC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BC-US-07
Record Dates: First submitted 2012-06-05; First posted 2013-08-15 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham Device (Sham Comparator): inactive AlphaCore device
  Interventions: Device: AlphaCore Device; Device: AlphaCore
- AlphaCore (Active Comparator): Active AlphaCore device
  Interventions: Device: AlphaCore Device; Device: AlphaCore

INTERVENTIONS:
Device: AlphaCore Device — Active stimulation to the vagal nerve
Device: AlphaCore — Active AlphaCore treatment

SUMMARY:
The purpose of this multi-center, prospective, double-blind, randomized, sham-controlled pilot study is to study feasibility and collect additional preliminary clinical data related to the safety and clinical benefits of non-invasive vagal nerve stimulation with the AlphaCore device for the treatment and prevention of exercise-induced bronchoconstriction, and to support the development and approval of a larger pivotal study.

The objectives of this study are (1) to gather preliminary safety and efficacy data of the AlphaCore device for the treatment of EIB (Treatment Visit 1) and prevention of EIB (Treatment Visit 2), (2) to validate the sham device (blinding effects, placebo effect) as an effective control for use in future clinical studies, and (3) to support the development and approval of a pivotal study, confirm data collection methods and endpoint definitions, and confirm appropriateness of the subject follow up plan.

DETAILED DESCRIPTION:
Study Design Summary Study Type: Prospective, randomized (allocated 1:1), double-blind, sham-controlled pilot study Sample Size: Up to 60 subjects Number of Sites: Up to 10 sites Anticipated Study Duration: 8 months

Number of Study Visits: Three:

1. Screening Visit
2. Treatment Visit 1 - treatment with AlphaCore (active or sham) after exercise challenge
3. Treatment Visit 2 - Prophylactic treatment with AlphaCore (active or sham) prior to exercise challenge

There will be a telephone follow-up call within 12-24 hours after the treatment visits occur as well as a 7-day (+/- 3 days) final phone call after Treatment Visit 2.

# of Study Arm(s): Two Arms

1. Active Treatment with the AlphaCore Device
2. Sham Treatment with an inactive sham device Blinding Double blind. The subject will be blinded to treatment assignment. Due to the treating Investigator's or designee designee's ability to detect differences in muscle effects between the active and sham device, the treating Investigator or designee cannot be blinded. Data assessors will be blinded.

ELIGIBILITY:
Inclusion Criteria:

1. Is able to give written Informed Consent.
2. Is between the ages of 18 and 60 years, male or female.
3. Has a history of breathlessness during and after exertion.
4. Normally controls or prevents EIB using a short acting beta-agonist (SABA).
5. Is willing to take a urine pregnancy test if female of childbearing potential and agrees not to become pregnant for the duration of the study.

Exclusion Criteria:

1. Has any condition that would prevent or otherwise inhibit reasonable exertion required to induce bronchoconstriction.
2. Is unable to perform acceptable-quality spirometry (FEV1 < 75% predicted).
3. Is currently using Beta2-adrenergic blockers (i.e. propranolol).
4. Has smoked within the past year, and/or more than 10 pack year history.
5. Has a history of lung cancer, chronic obstructive pulmonary disease (COPD), or other co-morbidity associated with irreversible narrowing of the airways.
6. Has an abscess or other infection or lesion (including lymphadenopathy) at the AlphaCore treatment site.
7. Has known or suspected moderate to severe atherosclerotic cardiovascular disease, carotid artery disease (e.g. bruits or history of TIA or CVA).
8. Has a clinically significant irregular heart rate or rhythm.
9. Has uncontrolled hypertension (systolic bp > 200 or diastolic bp >100), recent (within the last 3 months) heart attack, recent (within the last 3 months) stroke, known aortic aneurysm, or congestive heart failure (CHF).
10. Is currently implanted with an electrical and/or neurostimulator device, including but not limited to cardiac pacemaker, defibrillator, vagal neurostimulator, deep brain stimulator, spinal stimulator, bone growth stimulator, or cochlear implant.
11. Has a history of carotid endarterectomy, vagotomy (right or bilateral), dysaesthesia or vascular neck surgery on the right side.
12. Has been implanted with metal cervical spine hardware.
13. Has a recent or repeated history of syncope.
14. Has a recent or repeated history of seizures.
15. Has a condition that would interfere with VAS Dyspnea self-assessment.
16. Is pregnant or nursing, or of childbearing potential and is unwilling to use an accepted form of birth control.
17. Is participating in any other therapeutic clinical investigation or has participated in a clinical trial in the preceding 30 days.
18. Belongs to a vulnerable population or has any condition such that his or her ability to provide informed consent, comply with follow-up requirements, or provide self-assessments is compromised (e.g., homeless, developmentally disabled, prisoner).
19. Is an employee or relative of the Investigator or the clinical study site.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Weiman, Study Director — ElectroCore INC